CLINICAL TRIAL: NCT04200469
Title: Validation Of Quantitative Flow Ratio (QFR) - Derived Virtual Angioplasty
Acronym: QIMERA-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Carlos Baladron, PhD, Research Coordinator, Cardiology, Hospital Clínico Universitario de Valladolid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASVE-PI-19-1515
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Coronary Occlusion
Keywords: Quantitative Flow Ratio; QFR; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QFR Intervention (Experimental): Patients submitted to a coronary angiogram with at least one non-left main stable coronary stenosis between 50 and 90% and PCI indication with paired assessment of QFR, dFR, RFR and FFR, before and after PCI once informed consent is provided.
  Interventions: Diagnostic Test: Quantitative Flow Ratio (QFR) measurement

INTERVENTIONS:
Diagnostic Test: Quantitative Flow Ratio (QFR) measurement — Quantitative flow ratio (QFR) is a novel approach enabling rapid computation of FFR pullbacks from three-dimensional quantitative coronary angiography (3D-QCA) without using a pressure wire.

SUMMARY:
Prospective intervention study to assess the accuracy of the predicted QFR-derived virtual angioplasty compared to hyperaemic and non-hyperaemic pressure-wire derived indexes after PCI, as well as with QFR post-PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to a coronary angiogram with at least one non-left main stable coronary stenosis with PCI indication.

Exclusion Criteria:

* Severe stenosis of the left main coronary artery.
* Patients admitted with ST-elevation myocardial infarction.
* Culprit lesions in Non-ST-Elevation Acute Coronary Syndromes (NSTEACS) patients.
* Unability to identify the culprit lesion in NSTE-ACS patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Numerical agreement between predicted post PCI QFR (residual QFR) and post PCI dPR RFR-FFR, as well as direct QFR post-PCI mesurement. | 1 hour

SECONDARY OUTCOMES:
Sensitivity | 1 hour
Specificity | 1 hour
Summary of the receiver-operator characteristics curve (sROC) | 1 hour
Negative predictive value | 1 hour
Positive predictive value | 1 hour
Positive likelihood ratio | 1 hour
Negative likelihood ratio | 1 hour
Identification of independent predictors for increased predicted postPCI QFR (residual QFR) and post PCI dPR-RFR-FFR. | 1 hour

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Complejo Hospitalario Universitario, Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital de Lugo, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn JM, Park DW, Shin ES, Koo BK, Nam CW, Doh JH, Kim JH, Chae IH, Yoon JH, Her SH, Seung KB, Chung WY, Yoo SY, Lee JB, Choi SW, Park K, Hong TJ, Lee SY, Han M, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park SJ; IRIS-FFR Investigatorsdagger. Fractional Flow Reserve and Cardiac Events in Coronary Artery Disease: Data From a Prospective IRIS-FFR Registry (Interventional Cardiology Research Incooperation Society Fractional Flow Reserve). Circulation. 2017 Jun 6;135(23):2241-2251. doi: 10.1161/CIRCULATIONAHA.116.024433. Epub 2017 Mar 29. PMID 28356440
- [Background] Bech GJ, De Bruyne B, Bonnier HJ, Bartunek J, Wijns W, Peels K, Heyndrickx GR, Koolen JJ, Pijls NH. Long-term follow-up after deferral of percutaneous transluminal coronary angioplasty of intermediate stenosis on the basis of coronary pressure measurement. J Am Coll Cardiol. 1998 Mar 15;31(4):841-7. doi: 10.1016/s0735-1097(98)00050-3. PMID 9525557
- [Background] Bech GJ, De Bruyne B, Pijls NH, de Muinck ED, Hoorntje JC, Escaned J, Stella PR, Boersma E, Bartunek J, Koolen JJ, Wijns W. Fractional flow reserve to determine the appropriateness of angioplasty in moderate coronary stenosis: a randomized trial. Circulation. 2001 Jun 19;103(24):2928-34. doi: 10.1161/01.cir.103.24.2928. PMID 11413082
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Background] Adjedj J, De Bruyne B, Flore V, Di Gioia G, Ferrara A, Pellicano M, Toth GG, Bartunek J, Vanderheyden M, Heyndrickx GR, Wijns W, Barbato E. Significance of Intermediate Values of Fractional Flow Reserve in Patients With Coronary Artery Disease. Circulation. 2016 Feb 2;133(5):502-8. doi: 10.1161/CIRCULATIONAHA.115.018747. Epub 2016 Jan 5. PMID 26733607
- [Background] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Background] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Westra J, Tu S, Winther S, Nissen L, Vestergaard MB, Andersen BK, Holck EN, Fox Maule C, Johansen JK, Andreasen LN, Simonsen JK, Zhang Y, Kristensen SD, Maeng M, Kaltoft A, Terkelsen CJ, Krusell LR, Jakobsen L, Reiber JHC, Lassen JF, Bottcher M, Botker HE, Christiansen EH, Holm NR. Evaluation of Coronary Artery Stenosis by Quantitative Flow Ratio During Invasive Coronary Angiography: The WIFI II Study (Wire-Free Functional Imaging II). Circ Cardiovasc Imaging. 2018 Mar;11(3):e007107. doi: 10.1161/CIRCIMAGING.117.007107. PMID 29555835
- [Background] van Rosendael AR, Koning G, Dimitriu-Leen AC, Smit JM, Montero-Cabezas JM, van der Kley F, Jukema JW, Reiber JHC, Bax JJ, Scholte AJHA. Accuracy and reproducibility of fast fractional flow reserve computation from invasive coronary angiography. Int J Cardiovasc Imaging. 2017 Sep;33(9):1305-1312. doi: 10.1007/s10554-017-1190-3. Epub 2017 Jun 22. PMID 28642995
- [Background] Yazaki K, Otsuka M, Kataoka S, Kahata M, Kumagai A, Inoue K, Koganei H, Enta K, Ishii Y. Applicability of 3-Dimensional Quantitative Coronary Angiography-Derived Computed Fractional Flow Reserve for Intermediate Coronary Stenosis. Circ J. 2017 Jun 23;81(7):988-992. doi: 10.1253/circj.CJ-16-1261. Epub 2017 Mar 22. PMID 28331135
- [Background] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523
- [Background] Rimac G, Fearon WF, De Bruyne B, Ikeno F, Matsuo H, Piroth Z, Costerousse O, Bertrand OF. Clinical value of post-percutaneous coronary intervention fractional flow reserve value: A systematic review and meta-analysis. Am Heart J. 2017 Jan;183:1-9. doi: 10.1016/j.ahj.2016.10.005. Epub 2016 Oct 11. PMID 27979031
- [Background] Azzalini L, Poletti E, Demir OM, Ancona MB, Mangieri A, Giannini F, Carlino M, Chieffo A, Montorfano M, Colombo A, Latib A. Impact of Post-Percutaneous Coronary Intervention Fractional Flow Reserve Measurement on Procedural Management and Clinical Outcomes: The REPEAT-FFR Study. J Invasive Cardiol. 2019 Aug;31(8):229-234. Epub 2019 Jun 15. PMID 31199348
- [Background] Kikuta Y, Cook CM, Sharp ASP, Salinas P, Kawase Y, Shiono Y, Giavarini A, Nakayama M, De Rosa S, Sen S, Nijjer SS, Al-Lamee R, Petraco R, Malik IS, Mikhail GW, Kaprielian RR, Wijntjens GWM, Mori S, Hagikura A, Mates M, Mizuno A, Hellig F, Lee K, Janssens L, Horie K, Mohdnazri S, Herrera R, Krackhardt F, Yamawaki M, Davies J, Takebayashi H, Keeble T, Haruta S, Ribichini F, Indolfi C, Mayet J, Francis DP, Piek JJ, Di Mario C, Escaned J, Matsuo H, Davies JE. Pre-Angioplasty Instantaneous Wave-Free Ratio Pullback Predicts Hemodynamic Outcome In Humans With Coronary Artery Disease: Primary Results of the International Multicenter iFR GRADIENT Registry. JACC Cardiovasc Interv. 2018 Apr 23;11(8):757-767. doi: 10.1016/j.jcin.2018.03.005. PMID 29673507